CLINICAL TRIAL: NCT00684216
Title: Randomized Phase II/III Study of Second-line Endocrine Treatment Followed by Capecitabine Versus Capecitabine Followed by Endocrine Treatment in Patients With Metastatic Estrogen Receptor Positive Breast Cancer
Brief Title: Second-line Endocrine Treatment Followed by Capecitabine Versus Capecitabine Followed by Endocrine Treatment in Patients With Metastatic ER Positive Breast Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: acrual too slow
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: S. Rodenhuis, MD, NKI-AVL
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N07MAN; Eudract 2007-007030-20
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: metastatic; ER positive; PD during/after first line hormonal treatment
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; Tamoxifen; exemestane; Anastrozole; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): capecitabine followed by hormonal treatment
  Interventions: Drug: capecitabine; Drug: hormonal treatment (tamoxifen, exemestane, anastrozole or letrozole)
- 2 (Active Comparator): hormonal treatment followed by capecitabine
  Interventions: Drug: capecitabine; Drug: hormonal treatment (tamoxifen, exemestane, anastrozole or letrozole)

INTERVENTIONS:
Drug: capecitabine — 200 mg, BID, PO, QD until progression of disease
Drug: hormonal treatment (tamoxifen, exemestane, anastrozole or letrozole) — either tamoxifen or aromatase inhibitor (exemestane, anastrozole or letrozole), QD, until progression of disease

SUMMARY:
This trial studies the effects on quality of life and on time to second progression of the sequence endocrine therapy-capecitabine versus the sequence capecitabine-endocrine treatment. It is anticipated that the time on study (which is the time between randomization and the discontinuation of the second treatment in the sequence) will be similar for both arms of the study. The quality of life during this period, however, could be better in the patient group receiving the most effective first agent in the sequence. If this proves to be true, the conventional wisdom that endocrine therapy should be continued until no further endocrine options remain, must be abandoned.

DETAILED DESCRIPTION:
This is a randomized phase II/II study. Patients are randomized for the sequence capecitabine-hormonal therapy versus hormonal therapy- capecitabine. At progression the patient should receive the other protocol treatment (e.g. if the patient was randomized to capecitabine, at progression the treatment should be switched to hormonal treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Proven infiltrating breast cancer with distant metastases or inoperable locally advanced disease.
3. Positive estrogen receptor (≥ 10% positive nuclei at immunohistochemistry). Progesterone and HER-2 neu receptor have to be known.
4. - Progressive disease during first line hormonal therapy (either tamoxifen or aromatase inhibitor) for metastatic or inoperable locally advanced disease. Simultaneous use of LH-RH analogs is allowed. OR - Recurrence of disease (M1) during adjuvant hormonal therapy (either tamoxifen or aromatase inhibitor).
5. No prior chemotherapy for metastatic disease
6. Willing and able to participate in Quality of Life investigation -

Exclusion Criteria:

1. Other malignancy except carcinoma in situ, unless the other malignancy was treated 5 or more years ago with curative intent without the use of chemotherapy or radiation therapy.
2. Pregnancy or breast feeding women.
3. Contra-indications to the use of capecitabine
4. Known CNS metastases

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Quality of life during the study period: Physical functioning scale of the QLQ-C30; Global Health status/QoL of the QLQ-C30 | every 6 weeks

SECONDARY OUTCOMES:
Time to second progression and quality of life adjusted time to 2nd recurrence. | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Sjoerd Rodenhuis, MD, Principal Investigator — NKI-AvL
Locations (1):
- NKI-AVL, Amsterdam, Netherlands